CLINICAL TRIAL: NCT02023489
Title: Myocardial Lipid and Glycogen Metabolism & Cardiac Function in Patients With Impaired Glucose Tolerance or Type 2 Diabetes Mellitus and Calcium Sensing Receptor Mutations - A Cross Sectional Magnetic Resonance Spectroscopy and Imaging Study
Brief Title: Lipid and Glycogen Metabolism in Patients With Impaired Glucose Tolerance and Calcium Sensing Receptor Mutations
Acronym: RISC_7T
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Krebs, Prof. MD, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EK1128/2013
Record Dates: First submitted 2013-12-18; First posted 2013-12-30 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes Mellitus; Prediabetes (Insulin Resistance, Impaired Glucose Tolerance); Familiar Hypocalcuric Hypercalcemia; Healthy Volunteers; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Insulin Resistance; Glucose Intolerance; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Type 2 Diabetes Mellitus (Other)
  Interventions: Device: 1H/ 13C and 31P Magnetic Resonance Spectroscopy; Other: Hyperglycemic-hyperinsulinemic clamp
- Insulin sensitive volunteers (Other)
  Interventions: Device: 1H/ 13C and 31P Magnetic Resonance Spectroscopy; Other: Meal Tolerance Test; Other: Hyperglycemic-hyperinsulinemic clamp
- prediabetic subjects (Other)
  Interventions: Device: 1H/ 13C and 31P Magnetic Resonance Spectroscopy; Other: Meal Tolerance Test; Other: Hyperglycemic-hyperinsulinemic clamp
- familiar hypocalciuric hypercalcemic patients (Other)
  Interventions: Device: 1H/ 13C and 31P Magnetic Resonance Spectroscopy; Other: Meal Tolerance Test
- Type 1 diabetes mellitus (Other)
  Interventions: Device: 1H/ 13C and 31P Magnetic Resonance Spectroscopy

INTERVENTIONS:
Device: 1H/ 13C and 31P Magnetic Resonance Spectroscopy — Study participants will be studied in the fasting state after an overnight fast of at least 10 h. Participants will arrive at the MR-Centre in the morning of the study. Between 6:30 and 10:00 a.m., 1H MRI (3T) will be performed for the assessment abdominal adipose tissue distribution and composition as well as myocardial functional parameters. 1H/13C MRS examinations (7T) will be performed for measurements of myocardial, skeletal muscle and liver lipid content and composition as well as glycogen content. Additionally, ATP synthesis and energy metabolism will be assessed.
Other: Meal Tolerance Test — A meal tolerance test meal tolerance test according to Petersen et al. (PNAS, Vol 104, 2007) will be performed. After MRI and MRS examinations subjects will be returned at our outpatients clinic, where small polyethylene catheter will be inserted in an antecubital vein for hourly blood sampling. At 10:30 a.m. and 1:30 p.m. two liquid high carbohydrate meals of equal size containing all the required daily energy (30 kcal/kg of body weight; 55% carbohydrate, 10% protein, and 35% fat) with an additional 25% of the daily energy requirements added in the form of sucrose will be served.
  At 5 p.m. subjects will be returned at the MR - Centre for postprandial 1H / 13C MRS (7T) of muscle, liver and myocardial lipid and glycogen contents. Myocardial function parameters and abdominal fat distribution will be assessed again by 1H MRI (3T).
  Arms: Insulin sensitive volunteers; familiar hypocalciuric hypercalcemic patients; prediabetic subjects
Other: Hyperglycemic-hyperinsulinemic clamp — All volunteers will be admitted in the morning and basal 13C tracer enrichment will be assessed.
  At 8:00a.m. (0 min) a hyperglycemic-hyperinsulinemic-pancreatic clamp test will be initiated by somatostatin (-5-300 min: 0.1 µg·kg-1·min-1, UCB Pharma, Vienna, Austria) and insulin (0 - 8 min: 80 mU·min-1·m-2 body surface area; 8 -300 min: 40 mU·min-1·m-2 body surface area) infusion. Plasma glucose will be raised and maintained at ~180 mg·dL-1 by primed (0.2 g·kg-1)-variable dextrose infusion (20%w/v) enriched with [1-13C]glucose (40%w/w). A second catheter will be placed into an antecubital vein of the other arm and blood samples for the measurement of glucose, insulin and c-peptide. Glucose concentrations will be analysed immediately every 5 minutes, employing a glucose analyser. Myocardial glycogen concentrations will be measured before the clamp (-60 - 0 min) and from 90 min to 180 min during the clamp employing 13C MRS.
  Arms: Insulin sensitive volunteers; Type 2 Diabetes Mellitus; prediabetic subjects

SUMMARY:
Background:

Type 2 diabetes mellitus is a main risk factor for cardiovascular disease and heart failure, in part due to diabetic cardiomyopathy. However, the association between intracellular lipid accumulation and (myocardial) functional impairment is likely more complex than originally imagined. Recent studies suggest that not fat per se, but the content of saturated or unsaturated fatty acids might predict the development of cardiac steatosis and myocardial dysfunction.

In addition skeletal muscle and hepatic glycogen metabolism is impaired in patients with diabetes mellitus. Data from animal experiments suggest a relevant role of myocardial glycogen stores in ischemic preconditioning. Due to methodological limitations so far data on myocardial glycogen stores and myocardial lipid composition in humans are missing.

Hypothesis:

In addition to total ectopic lipid deposition in the myocardium, myocardial lipid composition, i.e. the relative abundance of saturated and unsaturated fatty acids, and impaired myocardial glycogen metabolism may play an important role in the development cardiac lipotoxicity leading to diabetic cardiomyopathy.

Pancreatic endocrine function and myocardial morphology and function is altered in patients with heterozygote inactivating mutations of the CaSR-gene / FHH.

Aims:

* Metabolic virtual biopsy of the myocardium for identification of specific patterns of intracellular lipid composition and myocardial glycogen metabolism as possible critical determinants of metabolic cardiomyopathy
* Characterization of the metabolic interplay between the myocardium, skeletal muscle, liver and adipose tissues in different stages of development of type 2 diabetes compared to patients with calcium sensing receptor mutation

Methods:

* 1H/13C and 31P magnetic resonance spectroscopy and imaging for measurements of myocardial, skeletal and liver lipid and glycogen content, abdominal adipose tissue distribution and composition, ATP synthesis and myocardial functional parameters
* Mixed meal tolerance tests to trace the postprandial partitioning of substrates between insulin sensitive tissues (myocardium, skeletal muscle, liver, adipose tissue).
* Hyperinsulinemic-hyperglycemic glucose clamp (HHC) with enrichment of the infused glucose with the stable isotope [1-13C]glucose to trace the incorporation of circulating glucose into myocardial glycogen

in healthy insulin sensitive volunteers, prediabetic insulin resistant volunteers with impaired glucose tolerance, healthy subjects, patients suffering from type 2 diabetes mellitus, patients suffering from type 1 diabetes and patients with heterozygote mutation in calcium sensing receptor.

DETAILED DESCRIPTION:
Background:

1. Type 2 diabetes mellitus is a main risk factor for cardiovascular disease and heart failure, in part due to diabetic cardiomyopathy. Ectopic intracellular lipid accumulation and impaired glycogen metabolism in skeletal muscle and liver and are closely associated with metabolic impairment in insulin resistant subjects and patients with diabetes mellitus. Recent evidence suggests that increased myocardial lipid accumulation might contribute to the development of myocardial dysfunction by direct toxic effects (lipotoxicity). However, the association between intracellular lipid accumulation and (myocardial) functional impairment is likely more complex than originally imagined. Recent studies suggest that not fat per se, but the content of saturated or unsaturated fatty acids might predict the development of cardiac steatosis and myocardial dysfunction.

   In addition carbohydrates stored as glycogen in muscle cells serve as readily available energy supply for contracting muscle. Skeletal muscle and hepatic glycogen metabolism is impaired in patients with diabetes mellitus. Data from animal experiments suggest a relevant role of myocardial glycogen stores in ischemic preconditioning. Due to methodological limitations so far data on myocardial glycogen stores and myocardial lipid composition in humans are missing.
2. Heterozygote inherited inactivating mutations in Calcium Sensing Receptor (CaSR)-gene leads to familiar hypocalciuric hypercalcemia (FHH), specified by mildly elevated plasma Ca and parathyroid hormone concentrations, whereas urine Ca excretion is inadequately low. However, in addition to the parathyroid gland CaSR is expressed in various tissues including the endocrine pancreas and the heart. So far it is unknown whether the endocrine function of the pancreas or myocardial morphology and/or function is altered in patients with FHH.
3. Altered hepatic energy metabolism might play an important role in the development of type 2 diabetes. Additionally, the lack of insulin delivery to the liver via the portal vein in type 1 diabetes might alter liver ATP synthesis. Therefore we aim to investigate hepatic energy metabolism non invasively with MRS.

Hypothesis:

In addition to total ectopic lipid deposition in the myocardium, myocardial lipid composition, i.e. the relative abundance of saturated and unsaturated fatty acids, and impaired myocardial glycogen metabolism may play an important role in the development cardiac lipotoxicity leading to diabetic cardiomyopathy.

Pancreatic endocrine function and myocardial morphology and function is altered in patients with heterozygote inactivating mutations of the CaSR-gene / FHH.

Hepatic and cardiac lipid and energy metabolism is altered in T1DM.

Aims:

* Metabolic virtual biopsy of the myocardium for identification of specific patterns of intracellular lipid composition and myocardial glycogen metabolism as possible critical determinants of metabolic cardiomyopathy
* Characterization of the metabolic interplay between the myocardium, skeletal muscle, liver and adipose tissues in different stages of development of type 2 diabetes compared to patients with calcium sensing receptor mutation

Methods:

* 1H/13C and 31P magnetic resonance spectroscopy (MRS) and imaging (MRI) for measurements of myocardial, skeletal and liver lipid and glycogen content, abdominal adipose tissue distribution and composition, ATP synthesis and myocardial functional parameters
* Mixed meal tolerance tests to trace the postprandial partitioning of substrates between insulin sensitive tissues (myocardium, skeletal muscle, liver, adipose tissue).
* Hyperinsulinemic-hyperglycemic glucose clamp (HHC) with enrichment of the infused glucose with the stable isotope [1-13C]glucose to trace the incorporation of circulating glucose into myocardial glycogen

in healthy insulin sensitive volunteers, prediabetic insulin resistant volunteers with impaired glucose tolerance, healthy subjects, patients suffering from type 2 diabetes mellitus, type 1 diabetes and patients with heterozygote mutation in calcium sensing receptor.

Relevance:

Despite intensive treatment of cardiovascular risk factors, heart diseases are still the main cause of death in diabetic patients. Thus, elucidation of mechanisms that link impaired lipid and/or glycogen metabolism and energy homeostasis to the development of heart failure appears to be crucial for the development of novel treatment strategies. Additionally, hepatic steatosis plays a challenging, emerging role in the treatment of liver disease, wherefore further insight in hepatic energy metabolism in various endocrine disease is urgently needed.

ELIGIBILITY:
Inclusion criteria for Type 2 DM patients:

* HbA1c: 7.0-8.0 %,
* m/f,
* age <90,
* no insulin therapy,
* normal liver function (transaminase <2 x than normal),
* no late diabetic complication (prolif. retinopathy, neuropathy, creatinin <1.5 mg/dl),
* female premenopausal patients: follicular = 1. phase of menstrual cycle,
* no evidence of coronary artery disease (ECG, patient history, symptoms).

Exclusion criteria for healthy controls:

* age <18 / >90a,
* dyslipidaemia (serum total cholesterol > 220 mg/dl, triglycerides > 150 mg/dl, LDL cholesterol > 130 mg/dl),
* arterial hypertension,
* cardiovascular diseases,
* thyroid disorders,
* bleeding disorders,
* medication potentially affecting glucose or lipid metabolism.

Inclusion criteria for the CaSR collective:

• genetically characterized heterozygote mutation in the CaSR gene

General exclusion criteria are:

* metal devices or other magnetic material in or on the subjects body which will be hazardous for NMR investigation [heart pacemaker, brain (aneurysm) clip, nerve stimulators, electrodes, ear implants, post coronary by-pass graft (epicardial pace wires), penile implants, colored contact lenses, patch to deliver medications through the skin, coiled spring intrauterine device, vascular filter for blood clots, orthodontic braces, shunt-spinal or ventricular, any metal implants (rods, joints, plates, pins, screws, nails, or clips), embolization coil, or any metal fragments or shrapnel in the body].
* BMI > 35 kg/m2
* tendency toward claustrophobia
* severe thyroid or liver disorders
* any acute illness within 2 weeks prior the study
* donation of blood within 30 days prior the study
* pregnancy
* malignancies, autoimmune disease
* AIDS, HIV, infectious hepatitis
* Plasma transaminases elevated > 3 fold
* Clinically relevant anemia
* Neurological disease
* Blood coagulation disorder
* severe dyslipidemia (serum triglycerides > 400 mg/dl, cholesterol > 300 mg/dl)
* arterial hypertension (RR > 180/100 mm Hg)
* clinical relevant cardiovascular diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
change in myocardial glycogen content | at baseline and during the third hour of the hyperglycemic clamp/ in the morning and at 5 p.m. after a meal tolerance test
  13C magnetic resonance spectroscopy for the assessment of myocardial glycogen content: Localized 13C NMR spectra will be obtained in a 7T Magnetom MR System (Siemens Healthcare, Erlangen Germany) with a dedicated butterfly-shaped 13C (15cm)/1H(21cm) transmitter/receiver coil (Stark Contrast, Erlangen, Germany) placed over or under the thorax. Recently introduced ISIS based or 1D CSI localization schemes will be applied. Absolute glycogen concentrations will be quantified by comparing the C1 glycogen peak (100.5 ppm) integral of tissue specific spectra with that of a glycogen standard taken under identical conditions. Corrections for loading of the coil and sensitive volume of the coil will be performed.

SECONDARY OUTCOMES:
change in myocardial lipid composition | at baseline and during the third hour of the hyperglycemic clamp/ in the morning and at 5 p.m. after a meal tolerance test
  Myocardial lipid measurements will be performed using localized 1H MRS. Anatomic imaging will be used to guide water suppressed Point RESolved Spectroscopy sequence (echo time, TE= 30 ms; minimal repetition time TR= 3 s; NS=64). The volume of the interest (VOI; approx. 6 - 8 cm3) will be placed over the interventricular septum. . An additional spectrum without water suppression (NS= 2x 4) will be used as internal reference. The spectra will be processed offline using AMARES time domain line fitting as implemented jMRUI software package. The myocardial lipid content will be determined from processed spectra as a ratio of the intensities of CH2 (1.25 ppm) and CH3 (0.8-0.9 ppm) group resonances to the intensity of the water resonance from non-water suppressed spectra of the same VOI.

OTHER OUTCOMES:
change in lipid content/composition in liver and skeletal muscle | at baseline and during the third hour of a hyperglycemic clamp/ in the morning and at 5:00 p.m. after a meal tolerance test
  Hepatic lipid content will be assessed using localized single voxel 1H MRS as published by our study-group. PRESS sequence (VOI= 3×3×3 cm3; TE= 30, 50, 70, 120 ms; NA= 4 for each TE) data acquisition will be performed during repetitive single breath holds. For intramyocellular lipid content STEAM sequence (VOI= 12x12x12 mm3; TE= 20 ms; TR= 4 sec, NA= 16) data acquisition will be performed in two volumes of interest positioned in soleus and tibialis anterior muscle.
  Lipid content will be calculated from ration of summed area of methylene and methyl resonance to that of water following the individual spin-spin relaxation correction as per cent of total tissue MRS signal (water + methylene + methyl).
differences in hepatic energy metabolism/ATP synthesis | baseline
  ATP synthesis will be assessed using 31P MRS. Patients with type 1 and type 2 diabetes, as well as pre diabetic insulin resistant subjects and insulin sensitive controls will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Michael Krebs, Prof MD, Principal Investigator — Medical University of Vienna, Department of Internal Medicine III, Division of Endocrinology and Metabolism
Locations (1):
- Medical University Of Vienna, Department of Internal Medicine III, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No